CLINICAL TRIAL: NCT03763565
Title: Effectiveness of HPV Vaccine Among Women Age Equal or More Than 20 Years
Brief Title: Effectiveness of HPV Vaccine in Thai Adult Women
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: National Vaccine Institute, Thailand (Other); Chulalongkorn University (Other); National Cancer Institute, Thailand (Other Government); Bumrungrad International Hospital (Other); Siriraj Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HPV 021; 2561.1/13 (Other Grant/Funding Number: National Vaccine Institute, Thailand)
Record Dates: First submitted 2018-12-03; First posted 2018-12-04 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Uterine Cervical Dysplasia; Papillomavirus Vaccines
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vaccinated group: Thai women who received at least one dose HPV vaccination at least 5 years ago, either by Bivalent or Quadrivalent HPV vaccines when they were 20-45 years old
  Interventions: Biological: Bivalent or Quadrivalent HPV vaccines
- Control group: Thai women who did not receive HPV vaccination, either by bivalent or quadrivalent HPV vaccine but have received Pap smear at their ages 20-45 years at least 5 years ago from the current enrollment time
  Interventions: Other: Control group

INTERVENTIONS:
Biological: Bivalent or Quadrivalent HPV vaccines — Vaccination with at least one dose of Bivalent or Quadrivalent HPV vaccines at least 5 years ago at the ages of 20-45 years
  Groups: Vaccinated group
Other: Control group — Thai women who did not receive HPV vaccination, either by bivalent or quadrivalent HPV vaccine but have received Pap smear at their ages 20-45 years at least 5 years ago from the current enrollment time
  Groups: Control group

SUMMARY:
* Background: The majority of the burden of HPV-related cervical cancer is in developing countries while most of the effectiveness reports of HPV vaccination are currently coming from developed countries. Also, currently many adult women are left without either HPV vaccination or cervical cancer screening. Effectiveness data of currently available HPV vaccines among adult women in developing countries are needed for women and healthcare workers and policy makers to best protect women from cervical cancer.
* Primary Study Objective:

  - To determine the effectiveness bivalent and quadrivalent HPV vaccines in reduction of cervical dysplasia (Low-grade Squamous Intraepithelial Lesion or worse; LSIL+) attributable to HPV types 16 or 18 after at least 5 years of vaccination among Thai women vaccinated at their ages 20-45 years with at least one dose of the HPV vaccine
* Secondary Study Objectives:

  * To measure the effectiveness of currently available bivalent and quadrivalent HPV vaccines in reducing the prevalence of HPV 16 or 18
  * To measure the effectiveness of HPV vaccines in reducing any abnormal Pap smear result (ASC-US+)
  * To compare the effectiveness of HPV vaccines according to the number of doses immunized
  * To find out risk factor(s) for HPV 16 or 18-related cervical dysplasia in this cohort
  * To assess the prevalence of other high-risk HPV types in vaccinated and non-vaccinated group
  * To determine direct and/or indirect cost of HPV vaccination
* The hypothesis to be tested: At least one dose of vaccination with bi- or quadri-valent HPV vaccine will reduce the prevalence of LSIL+ attributable to HPV 16/18 by 80% after at least 5 years of vaccination.
* Materials and Methods: This study will be a retrospective matched cohort study. Data is to be collected either by from samples for Pap and HPV test and/or HPV 16/18 genotyping of the recruited participants, or from existing medical records. HPV vaccinated women at their ages 20-45 years (vaccinated group) and women received Pap smear at their ages 20-45 years without vaccination (control group) will be included in the study. Pap smear and HPV test and/or HPV 16/18 typing result of 2 groups will be compared after ≥ 5 years of vaccination or baseline Pap smear. Those who don't have Pap smear results ≥ 5 years after vaccination or ≥ 5 years after the baseline Pap smear will be offered for a Pap smear and HPV 16/18 typing

ELIGIBILITY:
Inclusion Criteria

(vaccinated group)

* Thai women aged 20-45 years at the time of HPV vaccination
* Received at least 1 dose of bivalent or quadrivalent HPV vaccine at least 5 years ago
* Willing to provide written informed consent and receive Pap smear & HPV genotyping (only for those who need specimen collection for cervical cytology and HPV genotyping result)

(control group)

* Thai women without history of HPV vaccination
* Received Pap smear result at their ages 20-45 years at least 5 years ago
* Willing to provide written informed consent and receive Pap smear & HPV genotyping (only for those who need specimen collection for cervical cytology and HPV genotyping result)

Exclusion Criteria:

* Known pregnancy
* History of hysterectomy or excisional treatment of the cervix
* Known increased risk of bleeding
* Not willing to provide written informed consent

Ages: 25 Years to 53 Years | Sex: Female
Age Groups: Adult
Study Population: Vaccinated group: Thai women who received at least one dose of HPV vaccination, either by bivalent or quadrivalent HPV vaccine when they were 20-45 years old at least 5 years ago from the current enrollment time
  Control group: Women who did not receive any HPV vaccination, but received Pap smear result (conventional or liquid-based) when they were 20-45 years at least 5 years ago from the current enrollment time
Sampling Method: Non-Probability Sample
Enrollment: 993 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of Low-grade squamous intraepithelial lesion or worse (LSIL+) associated with HPV 16 or 18 | Sample collection in the project is single 1 day time for participants who received vaccination at least 5 years ago.
  LSIL or worse, including Atypical Glandular Cells, High-grade squamous intraepithelial lesion, Cervical intraepithelial neoplasia (CIN) grade 1-3, and cervical cancer which are associated with either HPV 16 or 18

SECONDARY OUTCOMES:
Cost-effectiveness of bivalent and quadrivalent HPV vaccination | Interview for direct and indirect cost survey will be single 1 day time for a participant.
  Direct and and indirect cost survey interview associated with HPV vaccination and its cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Punnee Pitisuttithum, Study Chair — Mahidol University
Locations (5):
- Thailand (5):
  - Bumrungrad International Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - National Cancer Institute, Thailand, Bangkok
  - Vaccine Trial Centre, Faculty of Tropical Medicine, Mahidol University,, Bangkok
  - Siriraj Hospital, Mahidol University, Bangkok